CLINICAL TRIAL: NCT00434629
Title: A Phase I Study of Bexxar® (Tositumomab and 131I-Tositumomab) Radioimmunotherapy in Patients With Relapsed or Residual CD20 Antigen-Expressing B-Cell Lymphomas Following Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Safety and Efficacy of Bexxar Therapy in the Treatment of Relapsed/Residual B-Cell Lymphoma After Autologous Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Stephen J. Schuster, MD, University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 18406; UPenn IRB#805353; GSK 106665
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: B-cell Lymphoma; Non-Hodgkin's Lymphoma
Keywords: lymphoma; Non-Hodgkin's lymphoma; B-cell lymphoma; Radioimmunotherapy; Bexxar; tositumomab; autologous hematopoietic stem cell transplantation
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma | interventions — tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bexxar — Day 0: Tositumomab, IV (in the vein) followed by test dose of 131I-Tositumomab, IV (in the vein) to determine treatment dose of 131I-Tositumomab.
  1-2 weeks after Day 0: Tositumomab, IV (in the vein) followed by therapeutic dose 131I-Tositumomab (in the vein).

SUMMARY:
Patients with B-cell lymphoma who relapse after autologous transplant tend to have a poor prognosis. Currently, there is no standard treatment for such patients. Bexxar is a radioactive antibody therapy that has shown a 60-80% response rate in non-transplanted patients with relapsed B-cell lymphoma. This study will test the safety and efficacy of Bexxar in the treatment of patients whose B-cell lymphoma has relapsed after an autologous transplant.

DETAILED DESCRIPTION:
High-dose chemotherapy followed by autologous stem cell transplantation (ASCT) has become the standard of care for relapsed/refractory chemotherapy-sensitive non-Hodgkin's lymphomas (NHL). However, one-half to two-thirds of such patients will relapse after ASCT, with subsequent poor prognosis, and new therapies are urgently needed for this patient population. Radioimmunotherapy (RIT) as a single agent therapy in patients with CD20 antigen-expressing relapsed or refractory low-grade, follicular, or transformed NHL has demonstrated overall response rates of 60-80% and has been approved by the FDA for use in this setting. While RIT is currently under investigation as a component of conditioning regimens for ASCT, the safety and efficacy of RIT after ASCT has not yet been well described. We will conduct a single-center Phase I dose-escalation trial of Bexxar (Tositumomab and 131I Tositumomab) for treatment of relapsed or residual CD20 antigen-expressing B-cell lymphomas following ASCT. Our primary aim will be to determine the safety, dose-limiting toxicity, and maximum tolerated dose of Bexxar in this post-ASCT patient population. Our secondary aim will be to describe the overall response rate, progression-free survival, time to treatment failure, and overall survival. Should Bexxar prove to be safe in this population, subsequent trials will be designed to investigate further the efficacy of RIT in the post-transplant setting.

ELIGIBILITY:
Inclusion Criteria:

* CD20 positive B-cell lymphoma
* Confirmed relapsed/refractory disease following autologous transplant
* Age ≤ 75 years
* Performance status 0 or 1
* Creatinine ≤ 1.5 or calculated creatinine clearance ≥ 60 ml/min
* Total bilirubin, AST, and ALT ≤ 1.5 x upper limit of normal (unless bilirubin due to Gilbert's)
* No active CNS disease
* No detectable bone marrow involvement by lymphoma on histopathologic bone marrow examination
* Bone marrow cellularity ≥ 15% on histopathologic bone marrow examination
* Availability of adequate stored autologous stem cell product (≥ 2 x 106 CD34+ cells/kg)

Exclusion Criteria:

* Active infection
* Pregnant woman are excluded from the study
* Subjects not using contraceptives are excluded from the study
* ANC ≤ 1,500/μL and/or platelet count ≤ 100,000/μL
* Life expectancy of ≤ 2 months
* Prior anti-B-cell radioimmunotherapy (e.g., Zevalin or Bexxar) [Patients who have received prior anti-B-cell monoclonal antibody therapy (e.g., rituximab or epratuzumab) will NOT be excluded.]
* Prior total body radiation therapy
* Positive human anti-mouse antibody (HAMA) testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
dose-limiting toxicity | Week 7 after Bexxar
maximum tolerated dose | Week 7 after Bexxar

SECONDARY OUTCOMES:
overall response rate | Week 13 after Bexxar
progression-free survival | 5 years after Bexxar
time to treatment failure | 5 years after Bexxar

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Schuster, MD, Principal Investigator — Abramson Cancer Center, University of Pennsylvania
Locations (1):
- Abramson Cancer Center, University of Pennsylvania, Philadelphia, Pennsylvania, United States